CLINICAL TRIAL: NCT04179747
Title: A Comparison of Psychotherapy and Pharmacotherapy in the Treatment of Erectile Dysfunction: A Pilot Study
Brief Title: Psychotherapy and Pharmacotherapy in the Treatment of Erectile Dysfunction: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University, Islamabad (Other)
Responsible Party: Principal Investigator, Ahmad Bilal, Principal Investigator, PhD Research Candidate, International Islamic University, Islamabad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 0925-0585
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Erectile Dysfunction
Keywords: Sexual Dysfunctions, Men Health
MeSH Terms: conditions — Erectile Dysfunction | interventions — Cognitive Behavioral Therapy; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The cognitive behavior psychotherapy was administered to participants in this treatment arm.
  Interventions: Behavioral: Cognitive Behavioral Psychotherapy
- Control Group (Active Comparator): This group received the administration of pharmacotherapy (PDE5i) for treatment of Erectile Dysfunction.
  Interventions: Drug: Sildenafil Citrate 50Mg Tab

INTERVENTIONS:
Behavioral: Cognitive Behavioral Psychotherapy — The Cognitive Behavior Psychotherapy was provided for a period of maximum 3 months.
  Other Names: Cognitive Behavior Psychotherapy
  Arms: Group A
Drug: Sildenafil Citrate 50Mg Tab — The participants in control group arm received Sildenafil Citrate 50mg tablet on demand for a period of maximum 3 months.
  Other Names: PDE5i
  Arms: Control Group

SUMMARY:
The study involved the administration of pharmacotherapy and cognitive behavior psychotherapy to individuals suffering from erectile dysfunction. The study was randomized controlled trial with two arms involving a control group. The study was conducted with an aim of pilot and feasibility study to evaluate the efficacy and suitability of cognitive behavior psychotherapy with individuals suffering from erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Men diagnosed with erectile dysfunction
2. Must be in the age range of 18 to 39 years
3. Must be in a stable heterosexual relationship
4. Must not be suffering from any medical or psychiatric illness

Exclusion Criteria:

1. Men not meeting criteria of diagnosis of erectile dysfunction
2. Men not in a heterosexual relationship
3. Men of or above the age of 40 years
4. Men diagnosed with any medical or psychiatric illness or obese men

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Functioning-5 | 3 months maximum
  The minimum scale score is 5. The maximum scale score is 25. The higher score indicates better erectile functioning.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale-21 | 3 months maximum
  The scale has three sub-scales.
  1. Depression sub scale, Minimum Score: Zero; Maximum Score: 42
  2. Anxiety sub scale, Minimum Score: Zero; Maximum Score: 42
  3. Stress sub scale, Minimum Score: Zero; Maximum Score: 42 The lowest scores on each of the sub scales indicate better functioning, the higher scores on each sub scale indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Bilal, MPhil, Principal Investigator — International Islamic University, Islamabad, Pakistan
Locations (1):
- Ahmad Bilal Private Practice, Chak Four Hundred Fifty-four, South Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilal A, Abbasi NUH. Development of an indigenous manual of cognitive behavior sex therapy for young men. J Family Med Prim Care. 2022 Aug;11(8):4127-4130. doi: 10.4103/jfmpc.jfmpc_1892_21. Epub 2022 Aug 30. PMID 36353027